CLINICAL TRIAL: NCT00792597
Title: Comparison of Three Methods of Hemoglobin Monitoring in Patients Undergoing Spine Revision or Hip Revision Surgery.
Brief Title: Comparison of Three Methods of Hemoglobin Monitoring
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 10-00524
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Blood Loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- spine or hip surgery

SUMMARY:
The purpose of this study is to compare the hemoglobin results obtained with 1) the HemoCue™, 2) the Masimo SpHb™, and 3) the UCSF Clinical Laboratory. The goal is to determine if these three values differ from each other during various levels of blood loss in the clinical care of patients for spine revision and hip revision surgery.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female 18 y/o or older
* American Society of Anesthesiology Classification 1, 2 or 3
* Scheduled to undergo spine or hip revision surgery

Exclusion Criteria:

* Pregnant or nursing
* Patients who in the study investigators clinical judgement would not be suitable for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
See description below | A minimum of three differences recorded during surgery
  Primary outcome is based on the difference between SpHb (Masimo SpHb™ continuous hemoglobin reading ) - tHb (laboratory hemoglobin determination).

SECONDARY OUTCOMES:
See description below | A minimum of three differences recorded during surgery
  Secondary outcome is based on the difference between a HemoCue™ derived hemoglobin determination - laboratory hemoglobin determination.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Miller, MD, Study Director — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Miller RD, Ward TA, Shiboski SC, Cohen NH. A comparison of three methods of hemoglobin monitoring in patients undergoing spine surgery. Anesth Analg. 2011 Apr;112(4):858-63. doi: 10.1213/ANE.0b013e31820eecd1. Epub 2011 Mar 8. PMID 21385985